CLINICAL TRIAL: NCT05294354
Title: Effects of Different Types of Acute Exercise on Cognitive Function: An Event-related Potential Study
Brief Title: Acute Exercise Type and Cognitive Function: An Event-related Potential Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yi-Ting Cheng, Graduate student, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PACNL_1100301_YTTY
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Exercise Training; Neurocognitive Function
Keywords: virtual reality; multi-domain exercise; executive function; inhibitory control
MeSH Terms: interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aerobic exercise group (AE) (Experimental): 35-min cycling at moderate intensity (50-60% heart rate reserve).
  Interventions: Behavioral: aerobic exercise group (AE)
- aerobic exercise with virtual reality group (AE-VR) (Experimental): 35-min cycling at moderate intensity (50-60% heart rate reserve) with 3D virtual reality.
  Interventions: Behavioral: aerobic exercise with virtual reality group (AE-VR)
- combined exercise group (CE) (Experimental): This 35-min exercise combines aerobic, bodyweight exercise, and meditation.
  Interventions: Behavioral: combined exercise group (CE)
- control group (Active Comparator): It has a 35-minute video about exercise science.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: aerobic exercise group (AE) — The participants will ride the cycle ergometer for 35 minutes. The training consisted of a 5-minute warm-up period followed by 25 minutes of moderate exercise and a 5-minute recovery.
  Arms: aerobic exercise group (AE)
Behavioral: aerobic exercise with virtual reality group (AE-VR) — The participants will receive the 3D VR training program and ride the cycle ergometer at the same time. The training protocol is similar to the aerobic exercise group.
  Arms: aerobic exercise with virtual reality group (AE-VR)
Behavioral: combined exercise group (CE) — The intervention consists of 5-minutes aerobic warm-up, 25-minutes bodyweight exercise, and 5-minutes mindfulness meditation for recovery. The participants will follow the video to do the program.
  Arms: combined exercise group (CE)
Behavioral: Control group — Participants will watch a 35-min video about exercise science.
  Arms: control group

SUMMARY:
This study aims to examine the effects of different types of acute exercise on cognitive functions in healthy adults.

DETAILED DESCRIPTION:
Acute exercise, a single session of exercise, has been shown to enhance cognitive functions. The meta-analysis research has suggested that such benefits might depend upon the types of exercise. However, the predominant types of exercise examined within this area of research are aerobic and resistance exercises. The effects of other types of exercises on cognitive functions are poorly understood. Accordingly, this study is going to examine the effects of different types of acute exercise [i.e., aerobic exercise (AE), aerobic exercise with virtual reality (AE-VR), and combined exercise (CE)] on cognitive functions.

140-180 healthy young adults will be recruited and then randomly assigned to the AE, AE-VR, CE, and Control groups for a 35-minute intervention. Cardiovascular fitness will be assessed beforehand. Additionally, Stroop tasks and several questionnaires will be conducted before and after the intervention. The targeted primary outcomes are changes in cognitive behavior performance (assessed by the Stroop tasks) and neuroelectrical indices (e.g., P3 of event-related potential). The secondary outcomes are the changes in exercise enjoyment, motivation, and emotion.

ELIGIBILITY:
Inclusion Criteria:

* no major psychiatric illness or physical disease
* able to do 30-minutes moderate exercise
* normal or corrected-to-normal vision
* right-handed
* moderate exercise ≤ 150 min/week

Exclusion Criteria:

* any neurological, respiratory, vascular, metabolic, or brain-relative disease
* any physical limitation or injury
* any wounds on the scalp
* have experience of using technology products
* regular engagement in exercise training programs

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Inhibition performance: Changes in Stroop test performance | 30 minutes each at the pretest and posttest
  The computerized Stroop test will be administrated to assess participants' cognitive functions, and their changes in reaction time and accuracy will be examined.
Changes in neuroelectrical activities | 30 minutes each at the pretest and posttest
  The neuroelectrical activities during the computerized cognitive tasks will be recorded. The changes in the event-related potential (e.g., P3) will be analyzed.

SECONDARY OUTCOMES:
Changes in physical activity enjoyment | 5-10 minutes each at the pretest and posttest
  The Chinese version of the physical activity enjoyment scale (PACES) questionnaire, with a total of 13 items, will be used to examine the changes in physical activity enjoyment. Participants will rate "how you feel at the moment about the exercise you have been doing" using a 7- point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it).
Changes in motivation | 3-5 minutes each at the pretest and posttest
  The Chinese version of the Motivation for Future Use questionnaire will be used. The scale consists of 3 items and each item is scored on a Likert-type scale that ranges from 1 to 7, with higher scores indicating a higher level of motivation.
Changes in emotion | 5-10 minutes each at the pretest and posttest
  The Chinese version of the positive and negative affect schedule (PANAS) will be used to assess the changes in emotion levels. It is a self-reporting questionnaire consisting of two 10-item scales and each item is scored on a Likert-type scale that ranges from 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Principal Investigator — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No